CLINICAL TRIAL: NCT04879212
Title: Clinical Effect of Electroacupuncture Combined With Fentanyl Patient-controlled Intravenous Analgesia on Postoperative Analgesia After Cesarean Section
Brief Title: Clinical Effect of Electroacupuncture on Postoperative Analgesia After Cesarean Sectionanalgesia After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-1029
Record Dates: First submitted 2021-04-18; First posted 2021-05-10 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2021-04

CONDITIONS: Cesarean Section
Keywords: Analgesia, Electroacupuncture
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: 1. PCIA +Acupuncture group
  2. PCIA +2 Hz Electroacupuncture group
  3. PCIA +20/100 Hz Electroacupuncture group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PCIA +Acupuncture group (Experimental): Acupuncturing bilateral Zusanli (ST36) and Sanyinjiao (SP6) to connect Huatuo brand electroacupuncture apparatus, but no electricity. Acupuncture was given once a day. PCIA（patient controlled intravenous analgesia）.
  Interventions: Other: PCIA +Acupuncture group:
- PCIA +2 Hz Electroacupuncture group (Experimental): Acupuncture bilateral Zusanli (ST36) and Sanyinjiao (SP6) to connect Huatuo brand electroacupuncture apparatus, and the ipsilateral Zusanli, Sanyinjiao were respectively connected as a loop. The parameters of electroacupuncture were set as 2Hz, continuous wave, 25min, and current intensity was 0.1-5.0mA. Acupuncture was given once a day.
  Interventions: Other: PCIA +Acupuncture group:
- PCIA +20/100 Hz Electroacupuncture group (Experimental): Acupuncture bilateral Zusanli (ST36) and Sanyinjiao (SP6) to connect Huatuo brand electroacupuncture apparatus, and the ipsilateral Zusanli, Sanyinjiao were respectively connected as a loop. The parameters of electroacupuncture were set as 20 / 100Hz, density wave, 25min, and current intensity was 0.1-5.0mA. Acupuncture was given once a day.
  Interventions: Other: PCIA +Acupuncture group:

INTERVENTIONS:
Other: PCIA +Acupuncture group: — Acupuncturing bilateral Zusanli (ST36) and Sanyinjiao (SP6)
  Other Names: PCIA +2 Hz Electroacupuncture group; PCIA +20/100 Hz Electroacupuncture group

SUMMARY:
Cesarean section is one of the most common operations in obstetrics. A survey shows that the rate of cesarean section in China is more than 40%, and even more than 70%. At present, the main analgesia methods after cesarean section are: patient controlled intravenous analgesia (PCIA), single injection of opioids into spinal canal, nerve block technique, combined or single oral drug for postoperative analgesia, etc. All kinds of postoperative analgesia methods have their own advantages and disadvantages. At present, PCIA is widely used in clinic, but it can cause side effects such as pruritus, nausea, vomiting and respiratory depression. Therefore, it is urgent to find a safe, effective, economic, reliable and operable treatment of PCIA for postoperative analgesia after cesarean section. Electroacupuncture is a technology combining traditional acupuncture and modern electrotherapy, which has a significant effect on acute and chronic pain. Studies have confirmed that electroacupuncture can help parturient women to deliver and relieve pain after delivery. However, there are few studies on the analgesic effect of Electroacupuncture on pain after cesarean section, and there are a few reports on wrist ankle acupuncture. On the basis of our previous research, we found that the frequency of 20 / 100Hz and 2Hz were the best for EA analgesia, and the density wave. Electroacupuncture is an ideal choice for PCIA analgesia after cesarean section because of its low price, rapid onset, long duration and no adverse drug reactions. "Zusanli" belongs to the stomach meridian of Foot Yangming. It is the meridian of multi Qi and multi blood. It has the effect of regulating meridians and collaterals, dredging Qi and blood, and treating various kinds of abdominal pain. Sanyinjiao belongs to the spleen meridian of foot Taiyin, which is the meeting of foot Taiyin, Jueyin and Shaoyin. Since ancient times, Sanyinjiao has been a commonly used acupoint to relieve labor pain. Modern studies have also shown that Sanyinjiao can relieve uterine contraction pain by relieving uterine smooth muscle spasm, improving the state of uterine ischemia and hypoxia, releasing a variety of central analgesic substances and so on Spleen and blood, liver tonifying and kidney tonifying. Therefore, on the basis of conventional PCIA analgesia combined with electroacupuncture at Zusanli and Sanyinjiao, we may play an auxiliary role in analgesia for puerpera after cesarean section.

DETAILED DESCRIPTION:
Electroacupuncture is an ideal choice for PCIA analgesia after cesarean section because of its low price, rapid onset, long duration and no adverse drug reactions. "Zusanli" belongs to the stomach meridian of Foot Yangming. It is the meridian of multi Qi and multi blood. It has the effect of regulating meridians and collaterals, dredging Qi and blood, and treating various kinds of abdominal pain. Sanyinjiao belongs to the spleen meridian of foot Taiyin, which is the meeting of foot Taiyin, Jueyin and Shaoyin. Since ancient times, Sanyinjiao has been a commonly used acupoint to relieve labor pain. Modern studies have also shown that Sanyinjiao can relieve uterine contraction pain by relieving uterine smooth muscle spasm, improving the state of uterine ischemia and hypoxia, releasing a variety of central analgesic substances and so on Spleen and blood, liver tonifying and kidney tonifying. Therefore, on the basis of conventional PCIA analgesia combined with electroacupuncture at Zusanli and Sanyinjiao, we may play an auxiliary role in analgesia for puerpera after cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Age 22-40 years old, gestational age 31-42 weeks;
* There was no electroacupuncture treatment before cesarean section;
* No food and drug allergy, no long-term use of analgesics; .They agreed and only participated in one clinical project and signed the informed consent form.

Exclusion Criteria:

* Suffering from complications after cesarean section, such as massive hemorrhage, etc;
* There was a history of chronic pain before operation;
* History of cognitive impairment;
* Skin lesions such as ulcers and eczema at the needling site are not suitable for needling;

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of times PCIA is used | 48 hours after operation
  Number of times PCIA is used

CONTACTS AND LOCATIONS:
Overall Officials: Ying Jin, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No